CLINICAL TRIAL: NCT06340009
Title: Comparison of Mime Therapy and Motor Imagery Technique on Facial Disability in Bell's Palsy.
Brief Title: MIME THERAPY vs MOTOR IMAGERY TECHNIQUE in Bell's Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01743
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Bell Palsy
MeSH Terms: conditions — Bell Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mime therapy group (Experimental): Mime therapy focuses on improving facial symmetry and muscle control through self-massage, breathing exercises, eye and lip closure exercises, letter and word exercises, and expression exercises in front of mirror
  Interventions: Other: mime therapy
- motor imagery group (Active Comparator): Motor imagery technique involves mental rehearsal of motor activities, activating similar brain regions as actual movements, which enhances neuroplasticity.
  Interventions: Other: motor imagery

INTERVENTIONS:
Other: mime therapy — 1. Facial Massage
  2. Frowning
  3. Close eyes
  4. Smile
  5. Fish Face
  6. Eyebrow raising
  7. Breathing exercise
  8. Blow cheeks
  9. Mouth opening and closing.
  10. Moving lips side to side
  11. Blow a candle.
  12. Nasal flaring
  13. Chewing exercise
  14. Rinse mouth
  15. Speaking vowels
  16. Fill mouth with water
  17. Fill rubber balloon
  18. Sucking water with straw
  Arms: Mime therapy group
Other: motor imagery — 1. Raising your eyebrows
  2. Showing angry face
  3. Closing and opening eyes
  4. Pouting
  5. Blowing cheeks
  6. Smiling
  7. Nasal flaring
  8. Blowing candle
  9. Deviating lips side to side
  10. Chewing something
  11. Speaking vowels
  Arms: motor imagery group

SUMMARY:
Bell's palsy, characterized by unilateral paralysis/paresis of facial muscles, is a condition with a significant impact on individuals' lives. It was first identified by scientist Sir Charles Bell, and its sudden onset can lead to social, psychological, and emotional distress. Left untreated, Bell's palsy can have long-lasting effects on a patient's quality of life, including loss of facial muscle control, emotional stress, and communication difficulties. Rehabilitation protocols encompass various physical therapy techniques, among which Mime therapy and Motor imagery technique have shown promise.

DETAILED DESCRIPTION:
While rehabilitation protocols have shown promise in enhancing facial muscle control, reducing disability, and preventing long-term complications, there remains a critical gap in the literature regarding the comparative effectiveness of various rehabilitation techniques. Currently, there is limited empirical evidence to guide healthcare professionals in selecting the most suitable rehabilitation approach for individual patients. The purpose of this study is to address this gap in knowledge by comparing two specific rehabilitation techniques: Mime therapy and Motor imagery technique. Understanding which of these rehabilitation techniques is more effective can significantly influence clinical practice and patient care. By conducting a systematic comparison, this study aims to provide evidence-based recommendations to healthcare professionals in selection of appropriate rehabilitation protocol for Bell's palsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40 years
* Both male and female
* Patients diagnosed with Bell's Palsy
* Paralysis/paresis of all muscle groups of one side of face

Exclusion Criteria:

* Patients diagnosed with facial palsy
* Patients with impaired cognition
* Patients diagnosed with other neurological diseases

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-08-22 (Estimated); Study Completion 2024-08-25 (Estimated)

PRIMARY OUTCOMES:
House-Brackmann Scale (HBS) | week 6
  A widely used scale to assess facial nerve dysfunction.Grades facial muscle function from I (normal) to VI (total paralysis). - Higher scores indicate more severe dysfunction.
Facial Disability Index (FDI) | week 6
  A patient-reported outcome measure assessing the impact of facial palsy on daily life.Assesses physical, social, and emotional functioning - Uses a questionnaire. - Higher scores indicate a greater impact on daily life.
Sunnybrook Facial Grading System | week 6
  An assessment tool for evaluating facial muscle function, including static and dynamic aspects.
Synkinesis Assessment Questionnaire (SAQ) | week 6
  An assessment tool specifically designed to evaluate synkinesis- related symptoms. Assesses the presence and severity of synkinesis symptoms during voluntary actions. - Uses a questionnaire. - Higher scores indicate more severe synkinesis-related symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Afridi, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Muzaffar Hospital, Sargodha, Pakistan

IPD SHARING:
Plan to Share IPD: No